CLINICAL TRIAL: NCT01978119
Title: A Randomised, Multi-Centre, Double-Blind, Double-Dummy, Two Way Cross-Over, Twelve Weeks Non-inferiority Study to Evaluate the Efficacy, Safety, and Tolerability of Combination Dry Powder of Fluticasone Propionate and Salmeterol 250/50 mcg Twice Daily Delivered Through a Capsule-Based Inhaler and a Multi-Dose Inhaler in Adults and Adolescents With Asthma
Brief Title: A Non-inferiority Study to Evaluate the Efficacy, Safety, and Tolerability of Combination Dry Powder of Fluticasone Propionate and Salmeterol (FSC) 250/50 Microgram (mcg) Twice Daily (BID) in Adults and Adolescents With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115645
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: Multi-Dose Inhaler; safety; Asthma; efficacy; pharmacodynamics; fluticasone propionate/salmeterol (FSC) 250/50 mcg; tolerability; Capsule-Based Inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects in this Arm will receive Regimen A followed by Regimen B. Regimen A: Placebo administered BID by Multi-Dose Inhaler followed by FSC (250/50 mcg) administered BID by Capsule-Based Inhaler. Regimen B: FSC (250/50 mcg) administered BID by Multi-Dose Inhaler followed by Placebo administered BID by Capsule-Based Inhaler
  Interventions: Drug: FSC; Drug: Placebo
- Sequence 2 (Experimental): Subjects in this Arm will receive Regimen B followed by Regimen A. Regimen B: FSC (250/50 mcg) administered BID by Multi-Dose Inhaler followed by Placebo administered BID by Capsule-Based Inhaler. Regimen A: Placebo administered BID by Multi-Dose Inhaler followed by FSC (250/50 mcg) administered BID by Capsule-Based Inhaler
  Interventions: Drug: FSC; Drug: Placebo

INTERVENTIONS:
Drug: FSC — Subject will be administered FSC 250 mcg/50 mcg via dry powder inhalation device or multi-dose dry powder inhalation device BID for each treatment period
Drug: Placebo — Subject will be administered placebo via dry powder inhalation device or multi-dose dry powder inhalation device BID for each treatment period

SUMMARY:
This is a multi-centre, randomised, double-blind, double-dummy, two way cross-over, 12 week non inferiority study to evaluate the efficacy, safety, and tolerability of FSC 250/50 mcg capsule-based inhaler and FSC 250/50 mcg multi-dose inhaler each administered BID in adults and adolescents with asthma. The primary objective of this study is to demonstrate that FSC 250/50 mcg administered BID by capsule-based inhaler is non-inferior compared to FSC 250/50 mcg administered BID by multi-dose inhaler . The study consists of six phases: Pre-screening, Screening/Run-in (3 weeks), Treatment Period 1 (12 weeks), Washout (minimum 3 weeks), Treatment Period 2 (12 weeks) and Follow-up (1 week). The total duration of the study for each subject will be at least 31 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >=12 and <=80 years of age at the time of signing the informed consent
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as premenopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone >40 milli international unit per milliliter (mIU/mL) and oestradiol <40 picogram (pg)/mL [<147 picomole per liter (pmol/L)] is confirmatory); Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study from Screening to follow-up contact) if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrolment. For most forms of HRT, at least 2 to 4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. After confirmation of their postmenopausal status, they can resume use of HRT during the study without use of a contraceptive method; child-bearing potential and is abstinent or agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) before the start of dosing to sufficiently minimise the risk of pregnancy at that point. Female subjects must agree to use contraception until at least 2 days post the last dose of study treatment; abstinence from penile-vaginal intercourse must be consistent with the preferred and usual lifestyle of the subject.
* Severity of disease: A best prebronchodilator FEV1 of >=40% to <=85% of the predicted normal value at Visit 1 (Screening and Run-in Visit). Predicted values will be based upon National Health and Nutrition Examination Survey (NHANES) III. If a subject is recorded as having Hispanic or Latino ethnicity, then the Mexican-American equations will be used (irrespective of race). If a subject is recorded as being of African-American/African heritage race, then the African American equations will be used. If a subject is recorded as being of Asian race, then the Asian adjustment will be used. Otherwise, the Caucasian equations will be used.
* Reversibility of disease: Demonstrated >=12% and >=200 mL reversibility of FEV1 within 10 to 40 minutes after 2 to 4 inhalations of salbutamol inhalation aerosol (or equivalent nebulised treatment with salbutamol solution) at Visit 1 (Screening and Run-in Visit).
* Current anti-asthma therapy: All subjects must be using an Inhaled Corticosteroid (ICS) with or without long-acting beta-adrenergic agonist (LABA) for at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit). Two populations are eligible for enrolment: - Subjects maintained on ICS monotherapy (FP 100 mcg to 250 mcg BID or equivalent) for at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit) or Subjects maintained on an ICS/LABA combination product (e.g., Fluticasone propionate/salmeterol 100/50 or 250/50 mcg BID or equivalent by other combination products or by separate inhalers) for at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit). Subjects taking budesonide/formoterol or beclomethasone/formoterol as needed must switch to budesonide/formoterol maintenance dosing (excluding the highest dose) with use of a SABA for symptom relief at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit). NOTE: Subjects on low dose ICS monotherapy should only be enrolled, if, in the opinion of the investigator, after review of their medical history and clinical examination, they will be able to benefit from both an increase in ICS dose and the addition of LABA therapy arising from and ICS/LABA combination.
* Ability to withhold LABA therapy: Other than what is provided during the study, LABA therapy is not permitted on the day of Visit 1 (Screening and Run-in Visit) and throughout the entire study. The last dose of LABA and LABA/ICS combinations are to be taken on the day before Visit 1. Sites should contact the medical monitor to discuss subject eligibility, for doses of commonly prescribed ICS and ICS/LABA combination medication; as mentioned in the study protocol.
* SABA: All subjects must be able to replace their current SABA treatment with rescue salbutamol/albuterol at Visit 1 (Screening and Run-in Visit) for use as needed for the duration of the study. Subjects must be able to withhold salbutamol/albuterol for at least 6 hours before each study visit.
* Liver safety criteria: Alanine aminotransferase (ALT) <=2 the upper limit of normal (ULN), Alkaline phosphatase and bilirubin <=1.5 ULN (isolated bilirubin >1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%) at Visit 1 (Screening and Run-in Visit).
* Electrocardiogram (ECG) safety criteria: The subject must have no ECG abnormalities that would, in the opinion of investigator, compromise subject safety, or significantly affect subject's ability to complete the trial. As such, the investigator will determine the clinical significance of any ECG abnormality and determine if a subject is precluded from entering the study. At Visit 1 (Screening and Run-in Visit), ECG safety criteria must be: QT interval corrected for heart rate (QTc) or QT interval corrected for heart rate according to Fridericia formula (QTcF) <450 msec or QTc <480 msec for subjects with bundle branch block; Investigators will be responsible for ensuring appropriate clinical interpretation of ECGs.
* The subject and/or the subject's legal guardian (if applicable) must be capable of giving informed consent/assent, which includes compliance with the study requirements and restrictions listed in the consent/assent form.

Exclusion Criteria:

* History of life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 10 years
* Respiratory infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 (Screening and Run-in Visit) and led to a change in asthma management, or in the opinion of the investigator, is expected to affect the subject's asthma status or ability to participate in the study
* Asthma exacerbation: Any asthma exacerbation requiring oral corticosteroids within 12 weeks of Visit 1 (Screening and Run-in Visit) or that resulted in overnight hospitalisation requiring additional treatment for asthma within 6 months before Visit 1 (Screening and Run-in Visit)
* Concurrent respiratory disease: A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma
* Other concurrent diseases/abnormalities: A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study. Additional excluded conditions/diseases are included in the study protocol
* Evidence of a severe exacerbation, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalisation or emergency department visit due to asthma that required systemic corticosteroids between Visit 1 (Screening and Run-in Visit) and Visit 2 (randomisation and Treatment Period 1 Baseline Visit)
* Oropharyngeal examination: A subject will not be eligible for the Run-in if he/she has clinical visual evidence of candidiasis at Visit 1 (Screening and Run-in Visit)
* Investigational medications: A subject must not have administered any investigational drug within 30 days before Visit 1(Screening and Run-in Visit) or within five half-lives of the prior investigational drug (whichever is the longer of the two). The prior investigational drug half-life may be confirmed with the prior investigational study sponsor or by consulting relevant study documentation
* Allergies: Drug allergy; Any adverse reaction including immediate or delayed hypersensitivity to any beta2 agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the FSC multi-dose inhaler and capsule-based inhaler (i.e., lactose), Milk protein allergy; History of severe milk protein allergy
* Concomitant medications: Administration of prescription or over the counter medication that would significantly affect the course of asthma, or interact with study treatment, such as: anticonvulsants (barbiturates, hydantoins, carbamazepine); polycyclic antidepressants; beta-adrenergic blocking agents; phenothiazines; and monoamine oxidase (MAO) inhibitors
* Immunosuppressive medications: A subject must not be using or require use of immunosuppressive medications during the study
* Cytochrome P450 3A4 (CYP3A4) inhibitors: Subjects who have received a potent CYP3A4 inhibitor within 4 weeks of Visit 1(Screening and Run-in Visit) (e.g., ritonavir, ketoconazole, itraconazole)
* Subject is unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) before the first dose of study treatment, unless in the opinion of the investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety
* Any subjects that have previously received or are currently receiving omalizumab
* Use of the excluded medications are included in the study protocol
* Compliance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, disease, or geographical location that seems likely (in the opinion of the investigator) to impair compliance with any aspect of this study protocol, including visit schedule and completion of the daily diaries
* Tobacco use: Current smoker or a smoking history of ≥10 pack-years (e.g., 20 cigarettes/day for 10 years). A subject must not have used inhaled tobacco products within the past 3 months (e.g., cigarettes, cigars or pipe tobacco). One pack year is defined as 20 manufactured cigarettes (1 pack) smoked per day for 1 year
* Pregnant females as determined by urine test at Visit 1 (Screening and Run-in Visit) or predosing. A confirmatory serum pregnancy test is required if the urine test is questionable or positive
* Lactating females
* A positive hepatitis B surface antigen or positive hepatitis C test result
* Subject is mentally or legally incapacitated
* Child in Care (CiC): A CiC is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a CiC can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The determination of whether a child meets the definition of CiC should be made with the study centre staff in consultation with the responsible institutional review board (IRB)/independent ethics committee (IEC).
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2015-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Russia (6):
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yaroslavl
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhia
  - GSK Investigational Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chan R, Sousa AR, Mallett S, Hynds P, Homayoun-Valiani F, Tabberer M, Mehta R. Assessment of the efficacy and safety of fluticasone propionate and salmeterol delivered as a combination dry powder via a capsule-based inhaler and a multi-dose inhaler in patients with asthma. Pulm Pharmacol Ther. 2016 Dec;41:19-24. doi: 10.1016/j.pupt.2016.09.002. Epub 2016 Sep 4. PMID 27599598
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 124 participants (par) were enrolled into the study, 33 participants were screen failures and 7 participants were run-in failures. A total of 84 participants were randomised and 82 participants were included in Intend to treat (ITT) population.
Groups:
- Sequence 1: Pl MD-DPI/FSC CB-DPI Then FSC MD-DPI/Pl CB-DPI: Participants self administered one inhalation of matching Placebo (Pl) via a multi-dose dry powder inhaler (MD DPI) and one inhalation of single capsule containing Fluticasone salmeterol combination (FSC) (250/50 microgram [mcg]) via a capsule-based unit dose (CB) DPI in the morning and evening in the Treatment Period 1 for 12 weeks. After washout period of 3 weeks participants self administered one inhalation of FSC (250/50 mcg) via the multi-dose DPI and one inhalation of of matching Placebo via the capsule-based unit dose DPI in the morning and evening in Treatment Period 2 for 12 weeks. Salbutamol/albuterol was provided to use as rescue medication.
- Sequence 2: FSC MD-DPI/Pl CB-DPI Then Pl MD-DPI/FSC CB-DPI: Participants self administered one inhalation of FSC (250/50 mcg) via a multi-dose DPI and one inhalation of Placebo via a capsule-based unit dose DPI in the morning and evening in Treatment Period 1 for 12 weeks. After washout period of 3 weeks participants self admnistered one inhalation of matching Placebo via a multi-dose DPI and one inhalation of FSC (250/50 mcg) via a capsule-based unit dose DPI in the morning and evening in Treatment Period 2 for 12 weeks. Salbutamol/albuterol was provided to use as rescue medication.
Period: Treatment Period 1 (12 Weeks)
Arm/Group | Sequence 1: Pl MD-DPI/FSC CB-DPI Then FSC MD-DPI/Pl CB-DPI | Sequence 2: FSC MD-DPI/Pl CB-DPI Then Pl MD-DPI/FSC CB-DPI
Started | 40 | 42
Completed | 38 | 42
Not Completed | 2 | 0
Not completed — Participants reached stopping criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout Period 1 (3 Weeks)
Arm/Group | Sequence 1: Pl MD-DPI/FSC CB-DPI Then FSC MD-DPI/Pl CB-DPI | Sequence 2: FSC MD-DPI/Pl CB-DPI Then Pl MD-DPI/FSC CB-DPI
Started | 38 | 42
Completed | 38 | 42
Not Completed | 0 | 0
Period: Treatment Period 2 (12 Weeks)
Arm/Group | Sequence 1: Pl MD-DPI/FSC CB-DPI Then FSC MD-DPI/Pl CB-DPI | Sequence 2: FSC MD-DPI/Pl CB-DPI Then Pl MD-DPI/FSC CB-DPI
Started | 38 | 42
Completed | 38 | 40
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants received one of the following 2 treatments in each of the two 12-week treatment periods separated by a 3-week washout period. One actuations of FSC (250/50 mcg) self administered twice daily (BID) (morning and evening) via multi-dose DPI plus one actuation of Placebo self administered BID (morning and evening) via capsule-based unit dose DPI or one actuation of Placebo self administered BID (morning and evening) via multi-dose DPI plus one actuation of FSC (250/50 mcg) self administered BID (morning and evening) via capsule-based unit dose DPI. Salbutamol/albuterol was provided to use as rescue medication.
Arm/Group | Overall Study
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 36
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 82

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Morning Forced Expiratory Volume in 1 Second (FEV1) at Day 85
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. The trough FEV1 is defined as morning prebronchodilator and predose (12 hours after the last evening dose Day 84). Trough FEV1 was measured electronically by spirometer in the morning, before using the bronchodilator and predose, at Week 12 (Day 85) of each Treatment Period. Baseline was defined as the value obtained predose (0 minutes) on day 1 in each treatment period. Change from Baseline within each period was calculated as trough FEV1 at Day 85 minus the period specific Baseline value. The change from Baseline in trough FEV1 was analysed using Mixed Model for Repeated Measures analysis, having fixed effect Participant level Baseline, Adjusted period-specific Baseline, Treatment group, Period, Visit, Visit by treatment, Visit by Participant level Baseline, Visit by Adjusted period-specific Baseline, with participant as a random effect.
Time Frame: Baseline and Day 85
Population: Intent-to-Treat (ITT) Population: all participants randomly assigned to treatment who received at least one dose of randomised study treatment in the Treatment Period. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- FSC Capsule-Based Unit Dose DPI: Participants received one actuation of Placebo self administered BID (morning and evening) via multi-dose DPI plus one actuation of FSC (250/50 mcg) self administered BID (morning and evening) via capsule-based unit dose DPI in either of two treatment periods for 12 weeks. Treatment periods were separated by washout period of 3 weeks. Salbutamol/albuterol was provided to use as rescue medication.
- FSC Multi-Dose DPI: Participants received one actuations of FSC (250/50 mcg) self administered BID (morning and evening) via multi-dose DPI plus one actuation of Placebo self administered BID (morning and evening) via capsule-based unit dose DPI in either of two treatment periods for 12 weeks. Treatment periods were separated by washout period of 3 weeks. Salbutamol/albuterol was provided to use as rescue medication.
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 78 | 80
Liter | 0.231 (0.0339) | 0.203 (0.0338)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Non-Inferiority or Equivalence — Non- inferiority was demonstrated if lower limit of the CI (0.025 one sided significance level) for the difference of the mean change from Baseline in trough FEV1 of FSC administered BID by capsule-based unit dose DPI versus FSC administered BID by multi-dose DPI is greater than -125 milliliter (mL); Repeated Measures Mixed Models; Mean Difference (Net) = 0.028, 95% CI 2-sided [-0.024 to 0.080]

2. Secondary Outcome: FEV1 Area Under the Curve From 0 to 12 Hours (AUC [0-12]) on Day 1 of Each Treatment Period
Description: The AUC was analysed using a mixed effects analysis of covariance (ANCOVA) with participant-level baseline (day 1 trough FEV1), adjusted period-specific baseline (day 1 trough FEV1), treatment group and period as fixed effects and participant as a random effect.
Time Frame: Day 1 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liter*hours
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 80 | 80
Liter*hours | 27.642 (0.3583) | 27.995 (0.3583)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Final Values) = -0.352, 95% CI 2-sided [-1.039 to 0.334]

3. Secondary Outcome: FEV1 AUC (0-12) at Day 85 of Each Treatment Period
Description: as for outcome 2
Time Frame: Day 85 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liter*hours
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 77 | 79
Liter*hours | 28.317 (0.4307) | 28.039 (0.4285)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Final Values) = 0.278, 95% CI 2-sided [-0.372 to 0.927]

4. Secondary Outcome: Change From Baseline in Morning Trough FEV1 at Day 28 and Day 56
Description: Pulmonary function was measured by FEV1, a measure of lung function, and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry at predose (Baseline), on Days 28 and 56 of each Treatment Period. Baseline was defined as the value obtained predose (0 minutes) on Day 1of each Treatment Period. Change from Baseline within each period was calculated as trough FEV1 at Day 28 and 56 minus the period specific Baseline value.The change from Baseline in trough FEV1 at Day 28 and Day 56 was analysed via the primary analysis model. Least Squares mean values for the change from Baseline in trough FEV1 at Day 28 and Day 56 were obtained from the primary analysis model (for each treatment and for the treatment difference), and displayed alongside corresponding 95% confidence intervals.
Time Frame: Baseline, Day 28, and Day 56
Population: ITT population, Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Participants at each time point may have been different therefore a total of 82 participants analyzed represents the overall ITT population.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 82 | 82
Liter
  Day 28, n=81, 80 | 0.245 (0.0402) | 0.238 (0.0405)
  Day 56, n=78, 80 | 0.224 (0.0378) | 0.202 (0.0377)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = 0.007, 95% CI 2-sided [-0.074 to 0.088] — Day 28 Change from Baseline Analysis
Statistical Analysis 2: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = 0.022, 95% CI [-0.049 to 0.092] — Day 56 Change from Baseline Analysis

5. Secondary Outcome: Change From Baseline (BL) in Morning Peak Expiratory Flow Rate (PEFR) Over 12 Weeks (From Paper Diary Card) for Each Treatment Period(TP)
Description: The PEFR is a paricipant's(par) maximum speed of expiration, as measured with a peak flow meter(PFM). All par were issued a PFM and instructed to perform the activity in triplicate in the morning prior to taking the bronchodilator. The best among the 3 readings was selected. Efficacy measurement was recorded by the par in the paper Diary Card for morning PEFR. The total PEFR over the 12 week TP was divided by the number of days with non-missing PEFR data to obtain an average for each par. Change from BL in average morning PEFR is the difference over 12 weeks for each TP compared to BL. BL is the average of the last 4 available recorded values during the last 7 days of the Screening Period (for TP 1) and of the Washout Period (for TP 2). The change from BL in the PEFR averaged over the 12-week TP was analysed using a mixed effects ANCOVA model with participant level BL PEFR, adjusted period-specific BL PEFR, treatment group, and period as fixed effects, and par as a random effect.
Time Frame: Baseline and up to Day 85 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 81 | 80
Liters per minute | 23.02 (3.325) | 18.67 (3.338)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = 4.35, 95% CI 2-sided [-1.34 to 10.05]

6. Secondary Outcome: Change From Baseline (BL) in Rescue Medication Use Over 12 Weeks (From Paper Diary Card) for Each Treatment Period (TP)
Description: Rescue medication usage for each 24-hour period is defined as the total numbers of puffs of Salbutamol/Albuterol within 24 hours (i.e. number taken during the day and number taken during the night). The total usage over the 12 week TP was divided by the number of days with nonmissing rescue medication data to get an average usage per participant. BL is the average of the last 4 available recorded values during the last 7 days of the Screening Period (for TP 1) and of the Washout Period (for TP 2). Change from BL in average usage of rescue medication was the difference over 12 weeks for each TP compared to BL. The change from BL in the percentage of rescue medication use averaged over the 12-week TP was analysed using mixed effects ANCOVA model, with par level BL rescue medication use, adjusted period-specific BL rescue medication use, treatment group and period as fixed effects and par as a random effect.
Time Frame: Baseline and up to Day 85 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 81 | 80
Puffs per day | -0.41 (0.086) | -0.36 (0.086)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.20 to 0.09]

7. Secondary Outcome: Change From Baseline in Day-time(AM) and Night-time (PM) Asthma Symptoms(Sy) From Paper Diary Card (PDC) Over 12 Weeks(wk) for Each Treatment Period(TP)
Description: AM Sy scores were recorded nightly on PDC using the scale:0=No Sy during day,1=Sy for one short period during day,2=Sy for two or more short periods during day,3=Sy for most of day-not affecting normal daily activities,4=Sy for most of day-did affect normal daily activities,5=Sy so severe-could not go to work or perform normal daily activities. Similarly, PM Sy scores were recorded every morning using the scale:0=No Sy during night,1=Sy causing me to wake once(or early),2=Sy causing me to wake twice or more(or early),3=Sy causing me to be awake most of night,4=Sy severe-did not sleep. BL= average of last 4 available of the last 7 days of Screening Period(TP 1) and of Washout Period(TP 2). Change from BL in average of daily scores=difference over 12 wks for each TP compared to BL. AM and PM Sy Scores were separately averaged over each of the two 12-wk TP. Total value of each endpoint over 12-wk TP was divided by number of days with non-missing data to obtain an average for each subject
Time Frame: Baseline and up to Day 85 of each Treatment Period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 82 | 82
Scores on the scale
  Day time (AM) score, n=81, 80 | -0.38 (0.685) | -0.25 (0.706)
  Night time (PM) score, n= 81, 80 | -0.16 (0.421) | -0.14 (0.389)

8. Secondary Outcome: Change From Baseline in the Percentage of Symptom-Free Days From Paper Diary Card Over 12 Weeks
Description: A Symptom-Free day was defined as a 24-hour period with no symptoms recorded. Percentage of Symptom-Free Days was calculated dividing number of Symptom-Free days by the length of the Treatment Period. The baseline value of change from baseline in % of symptom free days is defined as an average of the last 7 available recorded values the Screening Period (for treatment period 1) and of the Washout Period (for treatment period 2). Change from Baseline was the difference in percentage of Symptom-Free days at week 12 compared to Baseline. The change from Baseline in the percentage of Symptom-Free days averaged over the 12-week Treatment Period was analyzed, using mixed effects ANCOVA model, with participant level Baseline percentage of Symptom-Free days, adjusted period-specific Baseline percentage of Symptom-Free days, treatment group and period as fixed effects and participant as a random effect.
Time Frame: Baseline and up to Day 85 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free days
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 81 | 80
Percentage of symptom-free days | 11.36 (2.852) | 13.61 (2.864)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = -2.25, 95% CI 2-sided [-6.97 to 2.46]

9. Secondary Outcome: Change From Baseline in Asthma Control Test (ACT) Over 12 Weeks for Each Treatment Period
Description: The ACT is a 5-item questionnaire with a score of 1 to 5 for each item (1=poor control and 5=good control). The scores from each question were added to give an overall score. Baseline was defined as the value obtained predose (0 minutes) on day 1 of each Treatment Period. Change from Baseline was the difference in ACT score at the timepoint compared to Baseline score. The change from Baseline in overall ACT score was analysed, using mixed effects ANCOVA model, with participant level Baseline overall ACT score, adjusted period-specific Baseline overall ACT score, treatment group and period as fixed effects and participant as a random effect.
Time Frame: Baseline and up to Day 85 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Scores on the scale
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 78 | 80
Scores on the scale | 3.0 (0.35) | 3.2 (0.35)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.9 to 0.5]

10. Secondary Outcome: Change From Baseline in the Percentage (%) of Rescue-free Days Over 12 Weeks (From Paper Diary Card) for Each Treatment Period(TP)
Description: A rescue-free day is defined as a 24-hour period with no rescue medication usage recorded (i.e. both the day-time and night-time numbers of puffs of Salbutamol/Albuterol are zero). Percentage of Rescue-Free Days was calculated over each 12-week Treatment Period, dividing the number of rescue-free days by the length of the TP. The BL value of change from BL in % rescue free days is defined as an average of the last 7 available recorded values the Screening Period (for treatment period 1) and of the Washout Period (for treatment period 2). Change from BL was the difference over 12 weeks for each treatment period compared to BL. The change from BL in the % of rescue medication-free days averaged over the 12-week TP was analyzed, using mixed effects ANCOVA model, with par level BL % of rescue-free days, adjusted period-specific BL % of rescue-free days treatment group and period as fixed effects and par as a random effect.
Time Frame: Baseline and up to Day 85 of each Treatment Period
Population: ITT population, Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free days
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Number analyzed (Participants) | 81 | 80
Percentage of rescue-free days | 6.04 (2.391) | 6.81 (2.400)
Statistical Analysis 1: Comparison: FSC Capsule-Based Unit Dose DPI vs FSC Multi-Dose DPI; Test type: Superiority or Other; Mean Difference (Net) = -0.77, 95% CI 2-sided [-4.64 to 3.11]

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of administration of the study drug untill the follow-up contact (up to Week 28).
Description: SAEs and non-serious AEs were collected in members of the safety population, comprised of all participants randomised to treatment, who had received at least one dose of study medication.
Arm/Group | FSC Capsule-Based Unit Dose DPI | FSC Multi-Dose DPI
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 13/82 | 15/82
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC Capsule-Based Unit Dose DPI (N=82) | FSC Multi-Dose DPI (N=82)
Headache (Nervous system disorders) | 9 | 10
Hypertension (Vascular disorders) | 5 | 4
Blood pressure increased (Investigations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.